CLINICAL TRIAL: NCT02338544
Title: Application of Epiduo(R) PUMP in Daily Practice in Patients With Inflammatory Acne
Acronym: PUMP-it
Status: Completed | Type: Observational
Sponsor: Galderma Laboratorium GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: PUMP-it
Record Dates: First submitted 2015-01-12; First posted 2015-01-14 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene; Benzoyl Peroxide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 0.1% Adapalene / 2.5% Benzoyl peroxide — Epiduo® gel containing 0.1% adapalene + 2.5% benzoyl peroxide dispensed from a pump.
  Other Names: Epiduo(R) PUMP

SUMMARY:
The purpose of this observational trial is to assess application and convenience of Epiduo® PUMP under daily clinical practice conditions in patients with moderate to severe inflammatory acne.

DETAILED DESCRIPTION:
The objective of this observational trial is to assess application and convenience of Epiduo® PUMP under daily clinical practice conditions in patients with moderate to severe inflammatory acne using this drug in topical monotherapy or in combination with other drugs. In addition, efficacy of Epiduo® and incidence of adverse events will be assessed under marketed conditions. Also, patients' body beliefs will be recorded using the dysmorphic concern questionnaire.

The observational study is designed as a multicentre study, covering all parts of Germany. Participating investigators are dermatologists with an adequate patient pool of acne patients. The observation time per patient will up to 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥9 years
* The patient has been diagnosed with moderate to severe inflammatory acne (Leeds Grade 4-12)
* Chest/back affected allowed, but not required
* Topical therapy of acne with Epiduo® is indicated, the decision about treating the patient with Epiduo® has been made independently from this study

Exclusion Criteria:

* Pregnancy or breastfeeding
* Acne inversa
* Acne with preferential manisfestation of microcysts, macrocysts and macrocomedones
* Hypersensitivity to the medication or any of the ingredients
* Other contraindications mentioned in the Epiduo® SPC

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: About 2000 patients aged ≥9 years with moderate to severe inflammatory acne
Sampling Method: Probability Sample
Enrollment: 1388 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Severity of acne | at baseline and after up to 3 weeks of treatment
  Efficacy is assessed by change in severity of acne according to the Leeds revised grading system

SECONDARY OUTCOMES:
Patient-reported assessment | at follow-up
  Patient-reported assessment of application and convenience of Epiduo PUMP
Physician's assessment | at follow-up
  Overall assessment of Epiduo PUMP
Adherence | at follow-up
  Patient-reported frequency of the application
Dysmorphic concern | at baseline
  Assessment of patient's body beliefs using the dysmorphic concern questionnaire
Adverse drug reactions | at follow-up
  Documentation of adverse drug reactions

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Gieler, Prof. M.D., Principal Investigator — Universitätsklinikum Gießen und Marburg GmbH

IPD SHARING:
Plan to Share IPD: No